CLINICAL TRIAL: NCT05768191
Title: Comparative Efficacy of a Two Daily Mixed Insulin Injection Versus a Basal-bolus Scheme With Human Insulin in a Limited Resources Setting: a Multicenter Randomized Controlled Crossover Clinical Trial
Brief Title: Comparative Efficacy of a Two Daily Mixed Insulin Injection Versus a Basal-bolus Scheme With Human Insulin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Université NAZI BONI (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other); International Society for Pediatric and Adolescent Diabetes (Unknown); Société de Médecine Interne du Burkina Faso (Unknown); Association pour la Formation, la Recherche et l'Education sur le Diabète, Burkina Faso (Unknown)
Responsible Party: Principal Investigator, Yempabou Sagna, Principal Investigator, Université NAZI BONI
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2023-SOMIBF-01
Record Dates: First submitted 2023-03-01; First posted 2023-03-14 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin; Isophane Insulin, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Humulin N plus Humulin R (Active Comparator): 10 subjects will receive insulin human isophane suspension (Humulin N) twice daily plus regular human insulin (Humulin R) before meals
  Interventions: Drug: Humulin N plus Humulin R
- Premix human isophane suspension plus insulin human injection (Experimental): 10 subjects will receive premix insulin human isophane suspension and insulin human injection twice daily
  Interventions: Drug: premix insulin human isophane suspension and insulin human

INTERVENTIONS:
Drug: premix insulin human isophane suspension and insulin human — Sequence (Premix first, then Humulin N + Humulin R): Subjects randomized to this sequence will receive premix insulin, twice per day for 16 weeks. After the first 16 weeks, subjects will cross over to the Humulin N plus Humulin R sequence for a further treatment of 16 weeks
  Arms: Premix human isophane suspension plus insulin human injection
Drug: Humulin N plus Humulin R — Sequence (Humulin N + Humulin R first, then Premix): Subjects randomized to this sequence will receive basal bolus insulin scheme with Humulin N (twice daily) and Humulin R (before meals) for 16 weeks. After the first 16 weeks, subjects will cross over to the Premix sequence for a further treatment of 16 weeks
  Arms: Humulin N plus Humulin R

SUMMARY:
The goal of this clinical trial is to compare glycemic control and variability between children and adolescents with type 1 diabetes treated by a two daily injection of premixed human insulin (Humulin 30/70) and those who have a basal bolus scheme (Humulin N + Humulin R) in a resources limited setting.

The main question it aims to answer is: what is the effectiveness of premixed human insulin on glycemic control? Ten participants will be randomized initially to premix insulin human isophane suspension and insulin human injection (Humulin 30/70) twice daily, and 10 persons to insulin human isophane suspension (Humulin N) twice daily plus regular human insulin (Humulin R) before meals. At the end of the initial 16-wk treatment (period 1), all patients will be crossed over to the alternate treatment arm for an additional 16 wk (period 2). Insulin doses will be adjusted weekly by the clinical site according to a prespecified insulin intensification algorithm to achieve target fasting [<110 mg/dl (6.1 mmol/liter)], bedtime [<130 mg/dl (7.2 mmol/liter)], and premeal [<110 mg/dl (6.1 mmol/liter)] glucose levels until HbA1c was below 7.0%.

Subjects will receive training on the FreeStyle Libre CGMS System, electronic hand-held personal digital assistant (e-diary), and self-monitoring of blood glucose (SMBG), including recording glucose, insulin doses, and symptoms of hypo- or hyperglycemia.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 5 - 18 years of age
* Be diagnosed for at least 1 year at the date of inclusion.
* Have been regular at consultations during the last 12 years preceding inclusion (at least 3 visits)
* Willing and able to inject insulin human isophane and multi-day dosing of rapid acting human insulin.
* Willing and able to perform self-monitoring of blood glucose (SMBG) four times a day and continuous glucose monitoring (CGMS) for 48 hours at three time periods during the study
* Have (patient or guardian) a minimum 4 years primary school level
* Have (patient or guardian) a connected cellphone that can install the free FreeStyle link application and use connected messaging app

Exclusion Criteria:

* pregnant or lactating females
* opposition to participating in the study
* residing outside the towns where the care centers are located
* Any disease or condition (including abuse of illicit drugs, prescription medicines or alcohol) that in the opinion of the investigator or sponsor may interfere with the study compliance and completion of the study.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
To compare improvements from baseline in patient HbA1c when aggressively treated with insulin human isophane plus rapid acting human insulin vs treatment with Premix human insulin | 12 months

SECONDARY OUTCOMES:
frequency of hypo events (throughout the trial) | 8 months
  weekly frequency of hypo events and time below range
Quality of life score (baseline, week 32) (Using the Pediatric Quality of Life Inventory, 3.2 Diabetes module.) | 8 months
  The PedsQL 3.2 Diabetes Module is composed of 33 items comprising 5 dimensions for ages 8- 45 years and 32 items for ages 2-7 years. Items are reversed scored and linearly transformed to a 0-100 scale. Higher scores indicate lower problems
correlation between patient QoL and glucose variability as measured by CGMS (baseline, week 16 and week 32) | 8 months

CONTACTS AND LOCATIONS:
Locations (3):
- Burkina Faso (3):
  - CHU Souro Sanou, Bobo-Dioulasso, Houet
  - CHU de Tengandogo, Ouagadougou, Kadiogo
  - CHU Yalgado Ouedraogo, Ouagadougou, Kadiogo

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR